CLINICAL TRIAL: NCT07259265
Title: Longterm Outcomes of Vital and Non-vital Posterior Teeth Restored With Onlays and Single Crowns: a Randomized, Controlled, Clinical Trial
Brief Title: Vital and Non-vital Posterior Teeth Restored With Onlays and Single Crowns Using Three Different Restorative Materials.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. med. dent. Malin Strasding (Other)
Collaborators: Institut Straumann AG (Industry); Ivoclar Vivadent AG (Industry)
Responsible Party: Sponsor-Investigator, Dr. med. dent. Malin Strasding, PD Dr med dent, University of Geneva, Switzerland
Organization: University of Geneva, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GTC Study
Record Dates: First submitted 2024-12-19; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Decayed Teeth
Keywords: onlay; crown; partial coverage; full coverage; ceramic restoration
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crown restoration (Active Comparator): The tooth is restored with a conventional, full-coverage crown.
  Interventions: Procedure: Crown preparation
- Onlay restoration (Experimental): The tooth is restored with a defect-oriented onlay.
  Interventions: Procedure: Onlay preparation

INTERVENTIONS:
Procedure: Crown preparation — The conventional crown preparation will be performed.
  Arms: Crown restoration
Procedure: Onlay preparation — A defect-oriented tooth preparation is performed for an onlay restoration.
  Arms: Onlay restoration

SUMMARY:
The objective of this study is to assess the survival rate and the biological and technical outcomes of onlays and single crowns made out of different restorative materials on vital and non-vital teeth. The onlays are made either out of a lithium-disilicate glass ceramic (E.max CAD, Ivoclar Vivadent), hybrid ceramic (VITA ENAMIC, VITA Zahnfabrik) or out of a lithium aluminosilicate glass ceramic reinforced with lithium disilicate (N!ce, Straumann). The crowns are made either out of lithium aluminosilicate glass ceramic reinforced with lithium disilicate (N!ce, Straumann), hybrid ceramic (VITA ENAMIC, VITA Zahnfabrik) or lithium-disilicate glass ceramic (E.max CAD, Ivoclar Vivadent).

ELIGIBILITY:
Inclusion Criteria:

* • Subjects with the need for a fixed reconstruction in premolar and molar region with indication for either crown or onlay.

  * min. 18 years of age and ≤ 80 years
  * Patient with physical status PS1 and PS2 (according to Physical Status Classification System of the American Society of Anesthesiologists; Attachment 5)
  * Capable of providing written informed consent
  * Absence of any active periodontal and pulpal disease

Exclusion Criteria:

* Presence of conditions requiring chronic routine prophylactic use of antibiotics or prolonged use of steroids e.g. history of rheumatic heart disease, bacterial endocarditis, cardiac vascular anomalies, prosthetic joint replacements, etc.
* Patients with history of renal failure, bleeding disorders, metabolic bone disorder, uncontrolled endocrine disorders, HIV infection, Hepatitis
* History of neoplastic disease requiring the use of radiation or chemotherapy
* Inability to perform adequate oral hygiene
* Significant reduced saliva flow rate
* Unable or unwilling to cooperate for the trial period
* Allergy to any components of the reconstruction materials and cements
* Alcohol or drug abuse
* Pregnant or lactating women

Specific criteria:

* Root caries / root canal caries
* Extreme short dental arch (eSDA)
* Severe bruxism or clenching habits

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
Restoration survival | 5 years
  Survival of the inserted restorations

SECONDARY OUTCOMES:
Fractures of the restorations. | 5 years
  Any chipping (uncritical fractures) or critical fractures will be assessed.
Tooth vitality | 5 years
  The presence or absence of tooth vitality will be assessed by means of vitality test using cold spray.
Biological outcome - presence of secondary caries | 5 years
  Biological outcome - presence of secondary caries - of the treated teeth using magnification loops, a dental probe and radiographs.
Biological outcome - Bleeding on Probing | 5 years
  Bleeding on probing measures of the treated tooth using a periodontal probe.
Biological outcome - Plaque index | 5 years
  Assessment of the Plaque index of the treated tooth using a dental probe.
Biological outcome - tooth fractures | 5 years
  Assessment of tooth /root fractures using a dental probe and magnification loops.
Biological outcome - pocket probing depth | 5 years
  The pocket probing depth will be assessed in millimeters with a periodontal probe with 1mm distances.

OTHER OUTCOMES:
Restoration wear | 5 years
  Wear of the restorations by measuring the surface changes of the restorations over time. This is analyzed by means of digital intraoral scanning at different time points and measured in micrometers.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Geneva, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No
because of private patient data .